CLINICAL TRIAL: NCT03772704
Title: Multicenter Imaging in Lead Extraction Study
Acronym: MILES
Status: Completed | Type: Observational
Sponsor: The Cleveland Clinic (Other)
Collaborators: Philips Healthcare (Industry)
Responsible Party: Sponsor
Other Study IDs: 18-1480
Record Dates: First submitted 2018-12-07; First posted 2018-12-11 (Actual); Last update posted 2020-11-18 (Actual); Status verified 2020-11

CONDITIONS: Mechanical Complication of Cardiac Electronic Device

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 30 Days
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
The primary objectives of this registry is to correlate the amount of fibrosis as documented on Electrocardiogram (ECG) gated Computed Tomography (CT) scans with ease of advancing sheaths over the leads through the SVC zone during lead extraction.

DETAILED DESCRIPTION:
This is a multi-center, prospective, observational registry study which plans to enroll approximately 200 patients referred for Cardiac Implantable Electronic Device(CIED) lead extraction at one of the five study centers. The objective of this study is to determine whether a correlation exists between fibrosis detected on ECG gated cardiac CT and the ease of lead extraction as measured by need for extraction energy. All patients will be followed for 30 days post-lead extraction to assess vital status and re-hospitalizations via phone call

ELIGIBILITY:
Inclusion Criteria:

* Referred for CIED (Cardiac Implantable Electronic Device) lead extraction with at least 1 lead with dwell time greater than one year
* ≥ 18 years of age
* Appropriate candidate for chest/cardiac CT with contrast and full lead analysis

Exclusion Criteria:

* Atrial fibrillation with uncontrolled rate

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Referred patients for CIED lead extraction
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-12-13 (Actual); Primary Completion 2020-11-04 (Actual); Study Completion 2020-11-04 (Actual)

PRIMARY OUTCOMES:
Correlation of the presence and degree of fibrosis as determined by ECG gated cardiac CT with the presence and degree of fibrosis determined by ease of extraction sheath advancement | 30 days
  The presence and degree of fibrosis determined by the ease of extraction sheath advancement will be evaluated in three zones. Zone 1 will be the area before the Superior Vena Cava (SVC), Zone 2 in the SVC and Zone 3 after the SVC

SECONDARY OUTCOMES:
Percentage of ECG gated CT scans that show fibrosis | 30 days
  The percentage of ECG gated CT scans will be determined by scans that show little to no SVC (Zone 2) fibrosis, show little to no Zone 1 fibrosis, show little to no Zone 3 fibrosis, cardiac perforation, extravascular lead location
Major complications as defined by Heart Rhythm Society (HRS) 2017 consensus guidelines | 30 days
  major complications
Minor complications as defined by HRS 2017 consensus guidelines | 30 days
  minor complications
Mortality | 30 days
  Death assessed
Procedural outcomes | 30 days
  Operator ease of extraction (grade 1-5)
Fluoroscopy time | 30 days
  Fluoroscopy duration of time
Pathological reports from extracted leads | 30 days
  Pathology reports from extracted leads if available
Hospitalizations directly related to the extraction of leads or procedure related | 30 days
  Number of hospitalizations related to the extraction of leads or procedure related within 30 days post procedure

CONTACTS AND LOCATIONS:
Overall Officials: Bruce Wilkoff, MD, Principal Investigator — The Cleveland Clinic
Locations (5):
- United States (4):
  - United Heart and Vascular Clinic, Saint Paul, Minnesota
  - Northwell Health, Manhasset, New York
  - Duke University, Durham, North Carolina
  - Cleveland Clinic, Cleveland, Ohio
- Asklepios Klinik St. Georg, Hamburg, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Patel D, Vatterott P, Piccini J, Epstein LM, Hakmi S, Syed I, Koweek LM, Bolen M, Schoenhagen P, Tarakji KG, Francis N, Shao M, Wilkoff BL. Prospective Evaluation of the Correlation Between Gated Cardiac Computed Tomography Detected Vascular Fibrosis and Ease of Transvenous Lead Extraction. Circ Arrhythm Electrophysiol. 2022 Nov;15(11):e010779. doi: 10.1161/CIRCEP.121.010779. Epub 2022 Oct 28. PMID 36306341